CLINICAL TRIAL: NCT06147024
Title: Utilizing 3D Printed Personalized Aortic Lesion Models to Assist Surgeons in Preoperative Assessment and Planning of Aortic Aneurysm Surgery
Brief Title: Utilizing 3D Printed Personalized Aortic Lesion Models in Preoperative Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH112284
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Aortic Aneurysm
Keywords: 3D printing; pre-operative planning; thoracic aorta aneurysm; abdominal aorta aneurysm
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracic; Aortic Aneurysm, Abdominal | interventions — Historically Controlled Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- historical control group (Active Comparator): conventional preoperative assessment
  Interventions: Other: historical control
- 3D printed lesion model group (Experimental): using 3D printed lesion models for preoperative planning
  Interventions: Other: 3D printed lesion model

INTERVENTIONS:
Other: historical control — Received a conventional preoperative assessment
  Arms: historical control group
Other: 3D printed lesion model — Received 3D printed lesion models for preoperative planning
  Arms: 3D printed lesion model group

SUMMARY:
Using 3D printing technology to create personalized models of diseased heart and aortic blood vessels, surgeons can perform preoperative planning and evaluate relevant indicators.

DETAILED DESCRIPTION:
Background： Previous systematic reviews have indicated that approximately 82% of surgeries using 3D printed lesion models for preoperative planning have shown better surgical outcomes, and about half of the surgeries have demonstrated reduced operative time. In recent years, there have been numerous studies focusing on the application of 3D printing technology in aortic aneurysms. This study aims to employ 3D printing technology to fabricate personalized aortic blood vessel models with lesions.

Study Design： A single-centre, pilot study.

Methods： This study is a single-center, prospective clinical trial. The study plans to enroll 10 participants in the experimental group, and collect data from another 10 participants as the historical control group. The historical control group data will be matched-paired based on gender, age, and surgical type in sequential order.

Effect： We anticipate that through the use of 3D printed lesion models, we can reduce surgical time, decrease surgery-related complications, and enhance the smoothness of surgical team preparation for the procedure. Additionally, this approach can provide patients with a better understanding of their own condition and the upcoming surgical intervention.

Key words： 3D printing; pre-operative planning; thoracic aorta aneurysm; abdominal aorta aneurysm

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with thoracic or abdominal aortic aneurysm
* Signed surgical consent
* Non-emergent surgery
* Had 2D CT imaging within the last 6 months

Exclusion Criteria:

* Refusal to use lesion images for model creation
* Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-05 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
surgical time | immediately after the surgical procedure
  the duration of the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No